CLINICAL TRIAL: NCT05915468
Title: Large De-NOVo Coronary artEry Disease Treated With Sirolimus Drug Eluting Balloon: Prospective Evaluation of Safety & Efficacy of SELUTION SLR TM Drug Eluting Balloon (LOVE-DEB Registry)
Brief Title: Large De-NOVo Coronary artEry Disease Treated With Sirolimus Drug Eluting Balloon (LOVE DEB)
Status: Completed | Type: Observational
Sponsor: Wrightington, Wigan and Leigh NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: LOVE-DEB
Record Dates: First submitted 2022-12-06; First posted 2023-06-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this post-market Registry is to evaluate the safety and efficacy of SELUTION SLR, a Sirolimus Drug Eluting Balloon (DEB), in treating de novo native coronary artery disease in larger vessels (≥ 2.75 mm). This is a post-market registry that collects the data of patients who have been treated with a SELUTION DEB.

The primary objective is to evaluate the proportion of subjects who underwent Target Lesion Revascularization (TLR) within 1 year of the baseline PCI.

DETAILED DESCRIPTION:
This study is a prospective, observational, multicentre, single-arm registry designed to evaluate the clinical safety and performance of SELUTION SLR, Sirolimus-eluting balloon (SEB). The study population is made up of subjects who have undergone PCI using SELUTION DEB and are receiving standard of care (as per national guidelines). Subjects will be screened by site teams and offered the opportunity to participate in the registry after their procedure. Rationale for this study is to assess the safety and efficacy of SELUTION SLR, a sirolimus DEB, in larger vessels. The current evidence base for the safety & efficacy of sirolimus DEB in coronary vessels greater or equal 2.75mm is limited.

After an eligible subject has been treated with the SELUTION DEB, informed consent will be requested and the patient registered in the study. The study does not influence the choice of device utilised nor does it alter the routine standard of care.

Baseline data will be completed using medical notes and a baseline questionnaire will be completed by the subject. All recruited subjects will then be followed as per routine practice together with telephonic follow-up at 30 days and 12 months from the baseline PCI procedure date.

Potential subjects will be approached for informed consent after they have had a PCI procedure. They will be given the opportunity to ask any questions that they wish and given an appropriate amount of time to consider. Following registration, the baseline medical information will be collected from medical records and the subject will be asked to complete the SAQ-7 questionnaire.

The GP will be contacted to determine the survival status of the subject at 30 days (+/- 7 days) and 12 months (+/- 30 days) follow up, timed from date of baseline PCI. 30 day and 12 month follow up will done via the telephone and will consist of a verbally reported angina status assessment, recording of any adverse events, concomitant antiplatelet / anticoagulation medications and any interventional treatment that has occurred since previous contact. If the subject reports having angina at the 12 month time point then they will be asked to respond to the SAQ-7 questions over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients who have undergone PCI of at least one de-novo coronary lesion confirmed on coronary angiography using SELUTION SLR DEB, within 7 days prior to study registration.
* Vessel diameter must be ≥ 2.75 mm
* Bifurcation lesions: where main branch ≥ 2.75 mm and a DEB only strategy was applied in at least the main branch.
* Patients who give informed consent for participation in the study.

Exclusion Criteria:

* Patients with ST Elevation Myocardial Infarction (STEMI)
* Patients with cardiogenic shock.
* Patients who need urgent PCI following out of hospital cardiac arrest
* Patients with Left Main Stem or distal Left Main Stem bifurcation disease
* Patients with history of previous coronary revascularisation (PCI or CABG) prior to the baseline PCI
* Patients requiring calcium modification with rotational, orbital or laser atherectomy or intra-vascular lithotripsy (IVL)
* Patients with in-stent restenosis (ISR)
* Patients with Chronic Total Occlusions (CTO)
* Vessel diameter less than 2.75 mm
* Bifurcation lesion treated with stent (either main or side branch)
* Patients who have undergone cardiac transplant
* Patients with history of malignancy and life expectancy less than 12 months
* Patients who are pregnant or possibly pregnant.
* Patients have a known hypersensitivity or contraindication to Aspirin, Clopidogrel, Heparin or any other anticoagulation / antiplatelet therapy required for PCI, Sirolimus or contrast media.
* Patients scheduled to undergo elective surgery within 1-month post-index PCI.
* Patients who are currently participating in a clinical study of another drug or medical device and in whom assessment of the primary endpoint of that study has not been completed or clinically interferes with the endpoints of this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is made up of patients who have undergone PCI using SELUTION DEB and are receiving standard of care (as per national guidelines)
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Subject evaluation - Evaluate the proportion of subjects that underwent Target Lesion Revascularization (TLR) within 1 year of baseline PCI | 12 months
  Determined by percutaneous or surgical methods

SECONDARY OUTCOMES:
Patient reported recurrence of Angina | 12 months
  Assessed using the SAQ-7 questionnaire performed at baseline and via the telephone
All cause mortality | 12 months
  Cause of mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Wrightington Wigan & Leigh Teaching Hospitals NHS Foundation Trust, Wigan, United Kingdom

IPD SHARING:
Plan to Share IPD: No